CLINICAL TRIAL: NCT00012051
Title: A Randomised Phase III Study On The Effect Of The Chimeric Anti-CD20 Monoclonal Antibody (Mabthera) During Sequential Chemotherapy Followed By Autologous Stem Cell Transplantation In Patients With Relapse B-Cell Non-Hodgkin Lymphoma(HOVON 44 STUDY)
Brief Title: Chemotherapy and Peripheral Stem Cell Transplant With or Without Monoclonal Antibody Therapy in Treating Patients With Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Commissie Voor Klinisch Toegepast Onderzoek (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CKTO-2000-06; CDR0000068476 (Registry Identifier: PDQ (Physician Data Query)); HOVON-44; HOVON-44/CKVO-2000-06; EU-20042; ISRCTN95614846
Record Dates: First submitted 2001-03-03; First posted 2003-01-27 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2007-03

CONDITIONS: Lymphoma
Keywords: recurrent grade 3 follicular lymphoma; recurrent adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse | interventions — Filgrastim; Rituximab; Carmustine; Cisplatin; Cytarabine; Dexamethasone; Etoposide; Ifosfamide; Melphalan; Methotrexate; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Biological: rituximab
Drug: carmustine
Drug: cisplatin
Drug: cytarabine
Drug: dexamethasone
Drug: etoposide
Drug: ifosfamide
Drug: melphalan
Drug: methotrexate
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Peripheral stem cell transplant may be able to replace immune cells that were destroyed by the chemotherapy. Monoclonal antibodies, such as rituximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known if giving more than one drug (combination chemotherapy) plus peripheral stem cell transplant is more effective with or without monoclonal antibody therapy in treating non-Hodgkin's lymphoma.

PURPOSE: This randomized phase III trial is studying how well chemotherapy plus peripheral stem cell transplant with or without monoclonal antibody therapy works in treating patients with relapsed non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the partial and complete response rates in patients with relapsed, CD20 positive, aggressive B-cell non-Hodgkin's lymphoma treated with dexamethasone, cisplatin, and cytarabine in combination with etoposide, ifosfamide, and methotrexate with or without rituximab followed by carmustine, etoposide, cytarabine, melphalan, and autologous peripheral blood stem cell transplantation (APBSCT).
* Compare the effect of APBSCT with or without rituximab on the overall and event-free survival of these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive DHAP induction chemotherapy comprising dexamethasone orally or IV on days 1-4, cisplatin IV continuously over 24 hours on day 1, and cytarabine IV over 3 hours every 12 hours on day 2. Beginning 3-4 weeks after DHAP, patients receive VIM induction chemotherapy comprising etoposide IV over 2 hours on days 1, 3, and 5; ifosfamide IV over 1 hour on days 1-5; and methotrexate IV on days 1 and 5. Beginning 3-4 weeks after VIM, patients with partial or complete response after DHAP and VIM receive a second course of DHAP (patients with progressive or unresponsive disease after DHAP but responsive disease after VIM receive a second course of VIM) followed by filgrastim (G-CSF) subcutaneously beginning on day 10 and continuing until a target number of cells are collected.
* Arm II: Patients receive induction chemotherapy and G-CSF as in arm I. At 1 day after the last dose of each chemotherapy course, patients also receive rituximab IV once for a maximum of 3 courses.

At 4-5 weeks after the completion of the last induction chemotherapy course, responsive patients in both arms receive BEAM conditioning chemotherapy comprising carmustine IV over 60 minutes on day -6, etoposide IV over 60 minutes and cytarabine IV over 30 minutes on days -5 to -2, and melphalan IV over 15 minutes on day -1. Patients undergo autologous peripheral blood stem cell transplantation on day 0. After transplantation, patients in partial remission may undergo radiotherapy to nodal sites with residual tumor mass.

Patients are followed every 6 months for 3 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 296-340 patients (148-170 per treatment arm) will be accrued for this study within 4-5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed relapsed B-cell non-Hodgkin's lymphoma (NHL)

  * Diffuse large cell B-cell lymphoma
  * Grade III follicular center-cell lymphoma
  * Primary mediastinal B-cell lymphoma
* CD20 positive
* First relapse after doxorubicin containing regimen
* Documented remission of at least 3 months after first-line chemotherapy
* No Epstein-Barr virus post-transplantation lymphoproliferative disorder
* No CNS involvement

PATIENT CHARACTERISTICS:

Age:

* 18 to 65

Performance status:

* WHO 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* No hepatic dysfunction
* Bilirubin less than 2.5 times upper limit of normal (ULN)
* Transaminases less than 2.5 times ULN

Renal:

* No renal dysfunction
* Creatinine less than 2.0 mg/dL OR
* Creatinine clearance greater than 40 mL/min

Cardiovascular:

* No severe cardiac dysfunction
* No New York Heart association class II-IV heart disease

Pulmonary:

* No severe pulmonary dysfunction
* Vital capacity or diffusion capacity at least 70% predicted unless related to NHL involvement

Other:

* No active uncontrolled infection
* HIV negative
* No intolerance to exogenous protein administration

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 1 month since prior immunotherapy

Chemotherapy:

* See Disease Characteristics
* At least 1 month since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 1 month since prior radiotherapy

Surgery:

* Not specified

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2000-09; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Response rate
Event-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Edo Vellenga, MD, Study Chair — University Medical Center Groningen
Locations (17):
- U.Z. Gasthuisberg, Leuven, Belgium
- Netherlands (16):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Meander Medisch Centrum, Amersfoort
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Academisch Medisch Centrum at University of Amsterdam, Amsterdam
  - Medisch Spectrum Twente, Enschede
  - University Medical Center Groningen, Groningen
  - Medisch Centrum Leeuwarden - Zuid, Leeuwarden
  - Leiden University Medical Center, Leiden
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Sint Antonius Ziekenhuis, Nieuwegein
  - Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen
  - Daniel Den Hoed Cancer Center at Erasmus Medical Center, Rotterdam
  - HagaZiekenhuis - Locatie Leyenburg, The Hague
  - University Medical Center Utrecht, Utrecht
  - Isala Klinieken - locatie Sophia, Zwolle

REFERENCES:
- [Result] Vellenga E, van Putten WL, van 't Veer MB, Zijlstra JM, Fibbe WE, van Oers MH, Verdonck LF, Wijermans PW, van Imhoff GW, Lugtenburg PJ, Huijgens PC. Rituximab improves the treatment results of DHAP-VIM-DHAP and ASCT in relapsed/progressive aggressive CD20+ NHL: a prospective randomized HOVON trial. Blood. 2008 Jan 15;111(2):537-43. doi: 10.1182/blood-2007-08-108415. Epub 2007 Oct 30. PMID 17971487